CLINICAL TRIAL: NCT02788981
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase II Trial of Nanoparticle Albumin-Bound Paclitaxel (Nab-Paclitaxel, Abraxane®) With or Without Mifepristone for Advanced, Glucocorticoid Receptor-Positive, Triple-Negative Breast Cancer
Brief Title: Abraxane® With or Without Mifepristone for Advanced, Glucocorticoid Receptor-Positive, Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB16-0403
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Results first posted 2024-02-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer; advanced breast cancer; nab-paclitaxel; mifepristone; glucocorticoid receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Mifepristone; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nab-Paclitaxel+Mifepristone (Experimental): Patients will receive mifepristone 300 mg daily on the day prior to and day of each dose of nab-paclitaxel (100 mg/m2 on days 1, 8 and 15 of each 28 day cycle)
  Interventions: Drug: Mifepristone; Drug: Nab-Paclitaxel
- Nab-Paclitaxel+Placebo (Placebo Comparator): Patients will receive placebo and nab-paclitaxel (100 mg/m2 on days 1, 8 and 15 of each 28 day cycle)
  Interventions: Other: Placebo; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Mifepristone — Patients will receive mifepristone 300 mg daily on the day prior to and day of each dose of nab-paclitaxel (100 mg/m2 on days 1, 8 and 15 of each 28 day cycle).
  Other Names: KORLYM(R)
  Arms: Nab-Paclitaxel+Mifepristone
Other: Placebo — Patients will receive placebo and nab-paclitaxel (100 mg/m2 on days 1, 8 and 15 of each 28 day cycle).
  Arms: Nab-Paclitaxel+Placebo
Drug: Nab-Paclitaxel — Patients will either receive placebo and nab-paclitaxel (100 mg/m2 on days 1, 8 and 15 of each 28 day cycle) or patients will receive mifepristone 300 mg daily on the day prior to and day of each dose of nab-paclitaxel (100 mg/m2 on days 1, 8 and 15 of each 28 day cycle). Patients will receive mifepristone and nab-paclitaxel, or placebo and nab-paclitaxel. Not all three.
  Other Names: Abraxane®

SUMMARY:
This is a randomized, placebo-controlled, double-blind, phase II trial of nab-paclitaxel with or without mifepristone for advanced, glucocorticoid receptor-positive, triple-negative breast cancer. A total of 64 patients will receive nab-paclitaxel. Patients will be randomly assigned to either receive placebo or to receive mifepristone daily on the day prior to and day of each dose of nab-paclitaxel. Patients will be enrolled over 12 months and followed for 12 months following completion of study.

To expand and follow up on the investigators understanding of a potential pharmacokinetic (PK) interaction between nab-paclitaxel and mifepristone, investigators will perform PK studies in the first 20 patients enrolled at pre-specified "PK sites".

DETAILED DESCRIPTION:
Primary Objective:

To compare the progression free survival (PFS) of patients treated with nab-paclitaxel + placebo and patients treated with nab-paclitaxel + mifepristone.

Secondary Objectives:

1. To correlate percentage glucocorticoid receptor (GR) positivity in the most recent metastatic tumor biopsy (or in primary tumor if only primary tumor is available) with PFS in mifepristone and placebo groups.
2. To perform an exploratory assessment of overall response rate in both groups.
3. To collect information regarding overall survival in both treatment cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed breast cancer with stage IV or unresectable stage III disease.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. To be considered pathologically enlarged and measurable, a lymph node must be ≥15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm).
3. Triple-negative breast cancer (defined as estrogen receptor (ER) and progesterone receptor (PR) <10% positive; HER2 0-1+ by immuno-histochemistry (IHC) or fluorescence in situ hybridization (FISH) ratio <2.0)
4. Patients must have tumor block or slides available for testing, and tumor must be glucocorticoid receptor positive (defined as GR >10% moderate to strong staining by central lab). A formalin-fixed, paraffin-embedded surgical or core needle biopsy obtained from the primary tumor or from a metastasis and containing viable tumor tissue is required for this evaluation. Fine needle aspirates or other alternative cytology samples are not acceptable.
5. Patients may have received adjuvant chemotherapy and up to two prior chemotherapy for metastatic or locally recurrent disease. No prior nab-paclitaxel or mifepristone therapy for metastatic disease will be allowed.
6. Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of Nab-Paclitaxel in combination with Mifepristone in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
7. Eastern Cooperative Oncology Group performance status ≤ 2 (Karnofsky ≥ 60%).
8. Patients must have normal organ and marrow function as defined below

   * absolute neutrophil count >1,500 cells/mm3.
   * platelets ≥100,000/mcL
   * hemoglobin > 9.0 g/dL
   * total bilirubin< 1.5 mg/dL
   * alkaline phosphatase < 2.5 X upper limit of normal (ULN) or < 5 X ULN if bone mets are present
   * aspartate aminotransferase (AST) and Alanine transaminase (ALT) < 2.5 ULN or < 5 X ULN if liver mets are present
   * adequate renal function: creatinine ≤ institutional upper limit of normal OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
   * international normalized ratio (INR) < 1.5
9. Females of child-bearing potential (defined as a sexually mature woman who has not undergone hysterectomy, bilateral oophorectomy, or who has not been naturally postmenopausal for at least 24 consecutive months prior to study enrollment) must:

   * Commit to abstinence from heterosexual contact or agree to use effective contraception without interruption beginning at least 28 days prior to starting protocol therapy and while on study medication.
   * Have a negative serum pregnancy test result at screening and agree to ongoing pregnancy testing during the study dosing
10. Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following protocol discontinuation, even if he has undergone a successful vasectomy.
11. Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE).
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who are receiving any other investigational agents.
2. Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
3. Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
4. Patients with known brain metastases will be eligible as long as they have completed radiation to the brain, and have been off of corticosteroid therapy for at least 7 days.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to mifepristone or paclitaxel/nab-paclitaxel. Patients with a history of mild infusion reactions with paclitaxel who were able to continue to receive paclitaxel with corticosteroid premedication will be eligible to participate, as these cases were likely related to cremaphor and not paclitaxel.
6. Mifepristone can both inhibit CYP3A4 and induce CYP3A4. Addition of mifepristone to a pre-existing drug regimen may cause a mild and temporary increase in plasma drug concentration of drugs with significant CYP3A4 metabolism. Medications that are strong inducers of CYP3A4 such as carbamazepine, oxcarbazepine, phenobarbital, phenytoin, primidone, rifabutin, rifampin, rifapentine, St. John's Wort may decrease plasma mifepristone levels. Strong CYP3A4 inhibitor medications are expected to cause the largest increases in plasma mifepristone concentrations.

   Mifepristone may increase the plasma drug concentration of concomitant medications with metabolism mediated by CYP2C9/CYP2C8. Drugs with the largest increases will be those whose metabolism is largely or solely mediated by CYP2C9/2C8 and include: Non-steroidal Anti-inflammatory drugs (NSAIDs) and warfarin.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Pregnant women are excluded from this study because Mifepristone is an abortifacient agent with the potential for teratogenic effects.
9. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Mifepristone, breastfeeding should be discontinued if the mother wishes to participate in this study.
10. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Mifepristone. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
11. No history of long-term use of corticosteroids or concurrent short term use of corticosteroids is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nanda, M.D., Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - University of Chicago, Chicago, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo
Started | 13 | 16
Completed | 13 | 15
Not Completed | 0 | 1
Not completed — Patient chose to pursue alternative treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 49 (10) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 5 | 9 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Measured using the RECIST guideline v1.1
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo
Number analyzed (Participants) | 13 | 13
months | 3.0 [1.0 to 5.0] | 3.0 [1.0 to 6.0]

2. Secondary Outcome: Response Rate in Glucocorticoid Receptor (GR) Positivity
Description: Compare the response rate in GR positivity between the placebo and mifepristone groups using the RECIST guideline v1.1
Time Frame: 12 months
Population: Data on glucocorticoid receptor positivity was not collected.
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Response Rate
Description: Measured using the RECIST guideline v1.1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo
Number analyzed (Participants) | 13 | 13
Participants
  Responder | 3 | 5
  Non-Responder | 10 | 8

4. Secondary Outcome: Overall Survival
Description: Collected from date of randomization until death
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo
Number analyzed (Participants) | 13 | 14
months | 9.0 [6.0 to 28.0] | 6.0 [2.0 to 15.0]

ADVERSE EVENTS:
Time Frame: 24 months or until the subject is off study
Arm/Group | Nab-Paclitaxel+Mifepristone | Nab-Paclitaxel+Placebo
All-Cause Mortality (participants affected / at risk) | 12/13 | 14/15
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/15
Other Adverse Events (participants affected / at risk) | 13/13 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel+Mifepristone (N=13) | Nab-Paclitaxel+Placebo (N=15)
Fatigue (General disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel+Mifepristone (N=13) | Nab-Paclitaxel+Placebo (N=15)
Nausea (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Insomnia (Psychiatric disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 10
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 | 0
Neck stiffness (General disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 0
Flu like symptoms (General disorders) | 1 | 0
Peripheral edema (General disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Bladder spasms (Renal and urinary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Ocular edema (Eye disorders) | 1 | 0
Bilirubinemia (Investigations) | 1 | 0
Non-cardiac chest pains (General disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Extremity pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 6 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Investigations) | 6 | 1
Transaminitis (Investigations) | 1 | 2
Thrombocytopenia (Investigations) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was closed early, due to slow study accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT02788981/Prot_SAP_000.pdf